CLINICAL TRIAL: NCT06708559
Title: Immune Health Biomarkers and Fecal Microbiota in Filipino Breastfed Infants: A Prospective, Observational Study
Brief Title: Immune Health Biomarkers and Fecal Microbiota in Filipino Breastfed Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Asian Hospital and Medical Center, Muntinlupa City, Philippines (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2313INF
Record Dates: First submitted 2024-11-05; First posted 2024-11-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Immune system; Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Lactation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood & stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Breast-fed infants — Immune system characterization via blood and stool samples collection

SUMMARY:
This will be a prospective observational study aiming to investigate immune health biomarkers and fecal microbiota in 48-60 Filipino breastfed infants from birth to 12 months of age. An optional follow-up period of approximately 2 years will follow.

DETAILED DESCRIPTION:
This will be a prospective observational study in healthy term infants who are exclusively breastfed. Approximately 48-60 healthy breastfed infants aged ≥14 to ≤35 days at enrollment will be recruited and followed up until 12 month of age at 6 on-site visits: V1 (baseline), V3 (2 months), V5 (4 months), V6 (6 month), V7 (10months) and V8 (12 months).

The 12-month observational period will be followed by a 2year optional follow-up period for a total duration of the study of approximately 3 years.

The primary objective of this clinical study is to characterize early immune system development in breastfed Filipino infants by investigating infant blood markers of systemic immunity.

The secondary objectives will include the characterization of infant fecal markers of immune health and gut barrier function, infant blood and fecal microbiome, interactions between immune development and microbiome maturation, infant fecal metabolic profile and fecal pH, infant gastrointestinal (GI) tolerance, infant anthropometric measurements, infant complementary food intake as well as infant illness and infection.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained from parent(s)/ legally authorized representative(s) (LAR(s)).
2. Parent(s)/ LAR(s) must be able to provide evidence of parental authority and identity.
3. Parents/ LARs must understand the informed consent and other study documents.
4. Infants whose parent(s)/ LAR (s) has consented to blood collection as per protocol.
5. Able to temporarily store stool samples in a household freezer.
6. Infants whose parent(s)/LAR(s) are willing and able to comply with scheduled visits, and the requirements of the study protocol.
7. Infants whose parent(s)/LAR(s) can be contacted directly by telephone throughout the study.
8. Infants must meet all the following inclusion criteria to be eligible for enrollment into the study:

   1. Healthy term infant (≥37 weeks of gestation)
   2. At enrollment visit, postnatal age ≥14 to ≤35 days (date of birth = day 0)
   3. Birth weight is appropriate for gestational age (i.e., ≥ 2500g and ≤ 4500g)
   4. Infant has exclusively received breastmilk from birth to enrollment, and parent intends to continue exclusive breastmilk feeding until infant age 6 months.

Exclusion Criteria:

1. A medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   3. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study. Of note, children who are normally healthy but at the time of enrolment suffering from acute illness in a minor condition which are common in childhood and do not require some of the exclusionary medication mentioned below can be enrolled.
2. Presently receiving or have received prior to enrolment any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool microbiota and characteristics (e.g., oral, or systemic antibiotics, glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g., insulin or growth hormone); gastric acid secretion.
3. Infants whose parent(s) has(ve) not reached legal age of majority (18 years old) upon enrollment.
4. Currently participating or having participated in any interventional clinical trials since birth.

Ages: 14 Days to 35 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Approximately 60 healthy breastfed infants aged ≥14 to ≤35 days at enrollment. To ensure balanced sex representation of the study population, approximately 30 males and 30 females will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Markers of systemic immunity | Infant age ≥14 to ≤35 days, 2 months, 4 months, 6 months and 12months
  Descriptive statistics of plasma immune proteomics using mass cytometry or immunoassays, and vaccine-specific antibodies assessed by ELISA

SECONDARY OUTCOMES:
Fecal markers of immune health and gut barrier | Infant age ≥14 to ≤35 days, 2 months, 4 months, 6 months, 10 months and 12 months
  * Fecal markers of immune health and gut barrier, such as but not restricted to calprotectin and α-1-antitrypsin assessed by ELISA or alternative methods
  * Fecal cytokine profile using multiplex assays
Infant fecal microbiome | Infant age ≥14 to ≤35 days, 2 months, 4 months, 6 months, 10 months and 12months
  Microbiota composition, diversity, community types, and abundance of bacteria taxa
Fecal metabolic profile and pH | Infant age ≥14 to ≤35 days, 2 months, 4 months, 6 months, 10 months and 12 months
  pH and fecal organic acids, such as lactate, propionate, butyrate, acetate, valerate and total fecal organic acids, in wet stool weight and per dry stool weight
Plasma Metabolomics | Infant age ≥14 to ≤35 days, 2 months, 4 months, 6 months, and 12 months
  Untargeted Plasma metabolomics Analyses
GI Tolerance | Infant age ≥14 to ≤35 days, 1.5 months, 2 months, 3 months, 4 months, 6 months, 10 months and 12 months
  * Stool frequency and consistency, GI symptoms and GI-related behaviors collected via 1-day and 3-day GI Symptom and Behavior Diaries
  * GI burden score derived from the Infant Gastrointestinal Symptom Questionnaire (IGSQ-13)
Weight | Infant age ≥14 to ≤35 days, 1.5 months, 2 months, 3 months, 4 months, 6 months, 10 months and 12 months
  Measurement of weight in grams
Length | Infant age ≥14 to ≤35 days, 1.5 months, 2 months, 3 months, 4 months, 6 months, 10 months and 12 months
  Measurement of length in cm
Head circumference | Infant age ≥14 to ≤35 days, 1.5 months, 2 months, 3 months, 4 months, 6 months, 10 months and 12 months
  Measurement of head circumference in cm
Z-scores and percentiles | Infant age ≥14 to ≤35 days, 1.5 months, 2 months, 3 months, 4 months, 6 months, 10 months and 12 months.
  Changes in weight-for-age, weight-for-length, length-for-age, BMI-for-age, and head-circumference-for-age z-scores and percentiles calculated according to WHO standards
Infant illness and infection | Infant age 6 months
  Descriptive data and overall score derived from the Pediatric Immune System Index Questionnaire completed by parents
Infant Complementary Food Intake | Infant age 6-12months
  Descriptive data from complementary food questionnaire and 3-day food record
Long-term infant illness (during the optional follow-up) | Infant age 12 months, 18 months, 24 months, 30 months, and 36 months
  Descriptive data from the Infant Illness Questionnaire completed by parents

OTHER OUTCOMES:
Incidence of Adverse Events | From infant age ≥14 to ≤35 days to 12 months
  Incidents of adverse events from time of ICF signing at baseline, age ≥14 to ≤35 days, through the last study visit at age 12 months
Concomitant medications and treatments | From infant age ≥14 to ≤35 days to 12 months
  All concomitant medications / treatments (including type and duration) used to treat illnesses and other conditions will be recorded continuously from time of ICF signing at baseline, age ≥14 to ≤35 days, through the last study visit at age 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario JK Capeding, MD, Principal Investigator — Asian Hospital and Medical Center, Philippines
Locations (1):
- Asian Hospital and Medical Center, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No